CLINICAL TRIAL: NCT03245957
Title: HDL Dysfunction During the Acute Stage of Stroke
Acronym: RUSH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2016/CHU/06
Record Dates: First submitted 2017-08-08; First posted 2017-08-10 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ischemic stroke: Patients with ischemic stroke diagnosed by MRI or CT scan
  Interventions: Other: Ischemic stroke
- Haemorrhagic stroke: Patients without haemorrhagic stroke diagnosed by MRI or CT scan
  Interventions: Other: Haemorrhagic stroke
- Mimick stroke: Patients without haemorrhagic or ischemic stroke diagnosed by MRI or CT scan

INTERVENTIONS:
Other: Ischemic stroke — Patients with acute stage of stroke clinical picture, with ischemic, haemorrhagic or mimick stroke diagnosed using MRI or CT scan
  Groups: Ischemic stroke
Other: Haemorrhagic stroke — Patients with acute stage of stroke clinical picture, with ischemic, haemorrhagic or mimick stroke diagnosed using MRI or CT scan
  Groups: Haemorrhagic stroke

SUMMARY:
The study investigates the effect of plasma myeloperoxidase (MPO) concentrations on HDL dysfunction during the acute stage of ischemic and haemorrhagic strokes.

DETAILED DESCRIPTION:
MRI or CT scan are used to confirm the diagnosis of haemorrhagic, ischemic and mimick stroke.

Plasma anf HDL-MPO concentrations, as well as potent HDL dysfunction, are compared in the 3 cases.

The investigators hypothesis is that MPO concentrations and subsequent HDL dysfunction could be higher in ischemic strokes than in haemorrhagic ones. MPO could be a examined as a potent marker of early stage of ischemic stroke.

Plasma MPO levels could also be discriminant regarding the mimick strokes in patient exhibiting stroke clinical picture.

ELIGIBILITY:
Inclusion Criteria:

Patients with less than 12 hours stroke clinical signs:

* hemiparesis or hemiplegia
* unilateral sensitivity disorder
* language impairment
* balance disorder
* dizziness, bilateral or monocular vision totally or partially lost

Exclusion Criteria:

* Pregnancy
* head trauma since the last 3 months
* stroke since the last 3 months
* myocardial infarction since the last 3 months
* patient disagrees to be enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with clinical picture of early stage of stroke with the first signed lasting for less than 12 hours
Sampling Method: Non-Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2017-10-20 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Plasma MPO concentrations | Through study completion, an average of 6 hours
  Assessment of plasma MPO concentrations during acute stage of stroke

SECONDARY OUTCOMES:
HDL-MPO concentrations | Through study completion, an average of 6 hours
  Assessment of HDL-MPO concentrations during acute stage of stroke

OTHER OUTCOMES:
HDL dysfunction | Through study completion, an average of 6 hours
  Assessment of HDL function using inhibition test on cell culture

CONTACTS AND LOCATIONS:
Overall Officials: David COURET, MD, Principal Investigator — Centre Hpospitalier Universitaire de La REUNION
Locations (1):
- Chu Reunion Island, Saint-Pierre, Reunion Island, Reunion

IPD SHARING:
Plan to Share IPD: No